CLINICAL TRIAL: NCT03105609
Title: Enhancing the Lucentis (Ranibizumab) Management of Choroidal Neovascular Membranes With Hyperspectral Imaging
Status: Terminated | Type: Observational
Why Stopped: The delay between diagnosis and initiation of treatment was no longer consistent with standard of care
Sponsor: Center for Eye Research Australia (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Marc Sarossy, Dr, Center for Eye Research Australia
Other Study IDs: 16/1301H 21020
Record Dates: First submitted 2017-03-28; First posted 2017-04-10 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Macular Degeneration; Choroidal Neovascularization
Keywords: hyperspectral imaging, Ranibizumab
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Hyperspectral Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Naive wet age-related macular degeneration: Patients recruited to the study will be patients who meet the Australian MBS criteria for treatment of exudative CNV with Lucentis. For the duration of the study, the patients will have standard induction and monthly dosing of Lucentis (Ranibizumab; intravitreal; 0.5 mg) to allow comparison with published studies. The only extra intervention for the study is the acquisition of hyperspectral mages with the hyperspectral camera and the acquisition of additional fundus autofluorescence images to the clinical norm.
  Interventions: Device: Hyperspectral imaging

INTERVENTIONS:
Device: Hyperspectral imaging — Hyperspectral retinal images will be taken at baseline (before treatment with Lucentis) and then at 3 and 9 months after treatment.
  Other Names: Metabolic Hyperspectral Retinal Camera; Optina Diagnostics, Montreal, Canada

SUMMARY:
Clinical trial investigating the role of hyperspectral imaging in the management of patients undergoing standard clinical treatment for naive neovascular choroidal membranes in age-related macular degeneration.

DETAILED DESCRIPTION:
Observational trial of patients with choroidal neovascular membranes treated with Lucentis. Exploration and validation of a new form of retinal imaging called hyperspectral imaging.

Inclusion: Patients meet eligibility criteria other than FFA diagnosis and who are diagnosed with suspected exudative CNV on the OCT. (n=100 eyes) Procedure: Monthly doses of Lucentis. OCT scans will be taken prior to each injection. HSI image taken at baseline and at the 9-month time point.

Time frame: 6 months recruitment + 12 months follow-up + 6 months analysis.

All recruited patients will receive monthly doses of Lucentis as per the CMBS-approved protocol to allow comparison with other published studies. Lucentis will be administered in accordance with published standards of practice.

OCT scans will be taken prior to each injection. HSI image will be taken at baseline, three months and 9-month time points

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Willing to comply with all study procedures and be available for the duration of the study
* Male or female, aged 50-80
* In sufficiently good general health to be able to have a FFA
* CNV diagnosed by OCT
* Vision equal or better than 6/60 in the study eye
* No prior treatment in the study eye with anti-VEGF medication

Exclusion Criteria

* Significant media opacity.
* Known allergic reactions to components of the study product(s).
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 50-80 presenting for care in private ophthalmology practice with retinal specialists
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Hyperspectral image characteristics that predict response of choroidal neovascularisation to Lucentis | 3-9 months
  Hyperspectral images will be analysed to define specific characteristics that identify which types of choroidal neovascularisation will respond to Lucentis. Responsive patients will be differentiated from non-responders and distinguishing image features will be identified.

SECONDARY OUTCOMES:
Specific spectral signature for identification of exudative AMD | 3-9months
  Spectral bands of the HSI containing the most predictive information for diagnosis and treatment response will be characterised.

CONTACTS AND LOCATIONS:
Overall Officials: Marc G Sarossy, FRANZCO, Principal Investigator — Principal Investigator
Locations (1):
- Centre for Eye Research Australia, East Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
IPD not to be shared